CLINICAL TRIAL: NCT05171647
Title: A Randomized, Open-Label, Multicenter Phase III Study Evaluating Efficacy and Safety of Mosunetuzumab in Combination With Polatuzumab Vedotin in Comparison With Rituximab in Combination With Gemcitabine Plus Oxaliplatin in Participants With Relapsed or Refractory Aggressive B-Cell Non-Hodgkin's Lymphoma
Brief Title: A Study Evaluating Efficacy and Safety of Mosunetuzumab in Combination With Polatuzumab Vedotin Compared to Rituximab in Combination With Gemcitabine Plus Oxaliplatin in Participants With Relapsed or Refractory Aggressive B-Cell Non-Hodgkin's Lymphoma
Acronym: SUNMO
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO43643
Record Dates: First submitted 2021-12-06; First posted 2021-12-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — polatuzumab vedotin; tocilizumab; Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- M+P (Arm A) (Experimental): Participants will receive subcutaneous (SC) mosunetuzumab plus intravenous (IV) polatuzumab vedotin (M+P). Mosunetuzumab will be administered on Days 1, 8, and 15 of Cycle 1, and thereafter on Day 1 of Cycles 2-8. Polatuzumab vedotin will be administered on Day 1 of each cycle up to Cycle 6. Cycle length = 21 days.
  Interventions: Drug: Mosunetuzumab; Drug: Polatuzumab vedotin; Drug: Tocilizumab
- R-GemOx (Arm B) (Active Comparator): Participants will receive IV rituximab, IV gemcitabine, and IV oxaliplatin (R-GemOx) on Day 1 of each cycle for 8 cycles. Cycle length = 14 days.
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Mosunetuzumab — Participants will receive SC mosunetuzumab on Days 1, 8, and 15 of Cycle 1, and on Day 1 of Cycles 2-8 (cycle length = 21 days).
  Arms: M+P (Arm A)
Drug: Polatuzumab vedotin — Participants will receive IV polatuzumab vedotin every three weeks (Q3W) for 6 cycles (cycle length = 21 days).
  Arms: M+P (Arm A)
Drug: Tocilizumab — Participants will receive IV tocilizumab as needed to manage cytokine release syndrome (CRS) events.
  Arms: M+P (Arm A)
Drug: Rituximab — Participants will receive IV rituximab on Day 1 of each cycle for 8 cycles (cycle length = 14 days).
  Arms: R-GemOx (Arm B)
Drug: Gemcitabine — Participants will receive IV gemcitabine on Day 1 of each cycle for 8 cycles (cycle length = 14 days).
  Arms: R-GemOx (Arm B)
Drug: Oxaliplatin — Participants will receive IV oxaliplatin on Day 1 of each cycle for 8 cycles (cycle length = 14 days).
  Arms: R-GemOx (Arm B)

SUMMARY:
This study will assess the efficacy and safety of mosunetuzumab in combination with polatuzumab vedotin (M+P) in participants with relapsed or refractory (R/R) diffuse-large B-cell lymphoma (DLBCL), high-grade B-cell lymphoma, transformed follicular lymphoma (trFL) and FL Grade 3B (FL3B) in comparison with a commonly used regimen in this participant population, rituximab, gemcitabine and oxaliplatin (R-GemOx).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* CD20+ aggressive lymphoma as determined by the local hemopathology laboratory from the following diagnoses by 2016 World Health Organization classification of lymphoid neoplasms: DLBCL, not otherwise specified (NOS); high-grade B-cell lymphoma (NOS or double/triple hit); transformed follicular lymphoma; follicular lymphoma Grade 3b
* Have disease relapsed or refractory to at least one prior systemic therapy for aggressive non-Hodgkin's lymphoma (aNHL)
* Participants who have received only one prior line of therapy must be ineligible for autologous stem cell transplant (ASCT)
* Measurable disease
* Adequate hepatic, hematologic, and renal function
* Estimated creatinine clearance (CrCl) ≥ 30 mL/min by Cockroft-Gault method or other institutional standard methods
* Negative HIV test at screening. Participants with a positive HIV test at screening are eligible provided that, prior to enrollment, they are stable on anti-retroviral therapy for at least 4 weeks, have a CD4 count of at least 200 microliters, have an undetectable viral load, and have not had a history of opportunistic infection attributable to AIDS within the last 12 months

Exclusion Criteria:

* Pregnant or breast feeding, or intending to become pregnant during the study or within 3 months after the final dose of mosunetuzumab, 9 months after the final dose of polatuzumab vedotin, 12 months after the final dose of rituximab, 6 months after the final dose of gemcitabine, 9 months after the final dose of oxaliplatin, and 3 months after the final dose of tocilizumab, as applicable
* Inability to comply with protocol-mandated activity restrictions
* Prior treatment with mosunetuzumab or other CD-20-directed bispecific antibodies, or R-GemOx or Gem-Ox
* Prior treatment with polatuzumab vedotin, with the following exceptions: participants who have a documented response (partial response or complete response) to polatuzumab vedotin and an absence of PD within 12 months from the last dose of polatuzumab vedotin; participants who received up to 2 doses of a polatuzumab vedotin-containing regimen as bridging to CAR-T therapy, and either has a documented disease control (stable disease, partial response, or complete response), or were not assessed for response following treatment with polatuzumab vedotin
* Contraindication to any component of the study treatment
* Grade > 1 peripheral neuropathy
* Participants with Grade > 1 persistent toxicity related to prior anti-lymphoma treatment (except for alopecia and anorexia, or other toxicities not considered a safety risk for the participant per investigator's judgment)
* Received anti-lymphoma treatments with monoclonal antibodies, radio-immunoconjugates or antibody-drug conjugates (ADCs) within 4 weeks before the first dose of study treatment
* Treatment with any chemotherapeutic agent, or treatment with any other anti-lymphoma agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to the first dose of study treatment
* Treatment with radiotherapy within 2 weeks prior to the first dose of study treatment
* ASCT within 100 days prior to the first study treatment administration
* Prior treatment with chimeric antigen receptor (CAR) T cell therapy within 30 days before the first study treatment administration
* Prior allogenic stem cell transplant (SCT)
* Have had a solid organ transplantation
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* History of confirmed progressive multifocal leukoencephalopathy
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombination antibody-related fusion proteins)
* History of other malignancy that could affect compliance with the protocol or interpretation of results, with the exception of malignancies with a negligible risk of metastasis or death
* Currently have or have had a past history of central nervous system (CNS) involvement of lymphoma
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease. Participants with a history of stroke who have not experienced a stroke or transient ischemic attack in the past 2 years and have no residual neurologic deficits as judged by the investigator, or with a history of epilepsy who have had no seizures in the past 2 years while not receiving any anti-epileptic medications, are allowed
* Significant cardiovascular disease such as New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 6 months, unstable arrhythmias, or unstable angina
* Significant active pulmonary disease
* Participants with active symptoms of interstitial lung disease and/or pneumonitis, or those with a history of interstitial lung disease and/or pneumonitis within 6 months prior to the first dose of study treatment
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of the nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 2 weeks prior to the first study treatment administration
* Known or suspected chronic active Epstein-Barr virus (EBV) infection
* Recent major surgery within 4 weeks prior to the first study treatment administration
* Positive test results for chronic hepatitis B infection
* Acute or chronic hepatitis C virus (HCV) infection
* Have been administered a live, attenuated vaccine within 4 weeks before the first dose of study treatment administration or anticipation that such a live, attenuated vaccine will be required during the study
* Participants who have positive SARS-CoV-2 test within 7 days prior to enrollment (rapid antigen test result is acceptable)
* History of autoimmune disease
* Received investigational therapy, whether or not intended for lymphoma treatment, within 7 days prior to initiation of study treatment
* Clinically significant history of liver disease, including viral or other hepatitis, or cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the first occurrence of disease progression as determined by an independent review facility (IRF), or death due to any cause, whichever occurs first (up to 2.5 years)
Objective response rate (ORR) as determined by an independent review facility (IRF) | Up to 2.5 years

SECONDARY OUTCOMES:
ORR as determined by the investigator | Up to 2.5 years
Duration of response (DOR) | The time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as determined by the investigator and IRF (up to 2.5 years)
Overall survival (OS) | From randomization to death from any cause (up to 2.5 years)
PFS | From randomization to the first occurrence of disease progression as determined by the investigator, or death due to any cause, whichever occurs first (up to 2.5 years)
Complete response rate (CRR) | Up to 2.5 years
Duration of complete response (DOCR) | From the first occurrence of a documented complete response (CR) to disease progression or death from any cause, whichever occurs first, as determined by IRF and the investigator (up to 2.5 years)
Time to deterioration in physical functioning and fatigue as measured by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 | Up to 2.5 years
Time to deterioration in lymphoma symptoms as measured by the functional assessment of cancer therapy lymphoma subscale (FACT-Lym LymS) | Up to 2.5 years
Incidence of adverse events (AEs) | Up to 2.5 years
Change from baseline in peripheral neuropathy as measured by the functional assessment of cancer therapy/gynecologic oncology group - neurotoxicity (FACT/GOG-NTX) | Up to 2.5 years
Serum concentration of mosunetuzumab | Up to 2.5 years
Plasma concentration of polatuzumab vedotin | Up to 2.5 years
Change from baseline in the EuroQol 5-dimension, 5-level questionnaire (EuroQol EQ 5D-5L) index-based scores | Up to 2.5 years
Change from baseline in the EuroQol EQ 5D-5L visual analog scale (VAS) scores | Up to 2.5 years
Incidence of anti-drug antibodies (ADAs) to mosunetuzumab | Up to 2.5 years
Incidence of anti-drug antibodies (ADAs) to polatuzumab vedotin | Up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (52):
- United States (4):
  - City of Hope Cancer Center, Duarte, California
  - St. Luke's Hospital, Chesterfield, Missouri
  - Ascension Seton Infusion Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Argentina (4):
  - Hospital Aleman, Buenos Aires
  - Instituto Alexander Fleming, Buenos Aires
  - FUNDALEU, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
- Brazil (5):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clínicas FMRP-USP, Ribeirão Preto, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
  - D'or Instituto de Pesquisa e Educação, São Paulo
- Canada (3):
  - Hamilton Health Sciences - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Chum Hopital Notre Dame, Montreal, Quebec
- China (6):
  - Sichuan Cancer Hospital, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - Cancer Center, Sun Yat-sen University of Medical Sciences, Guangzhou
  - Tianjin Cancer Hospital, Tianjin
  - Tongji Hosp, Tongji Med. Col, Huazhong Univ. of Sci. & Tech, Wuhan
  - Henan Cancer Hospital, Zhengzhou
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Ichilov Sourasky Medical Center, Tel Aviv
- Japan (6):
  - Kyushu University Hospital, Fukuoka
  - Hokkaido University Hospital, Hokkaido
  - Tohoku University Hospital, Miyagi
  - Kindai University Hospital, Osaka
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Yamagata University Hospital, Yamagata
- Mexico (5):
  - Health Pharma Professional Research, Mexico City, Mexico CITY (federal District)
  - Superare Centro de Infusion S.A. de C.V., Mexico City, Mexico CITY (federal District)
  - Hospital Universitario Dr. Jose E. Gonzalez, Monterrey, Nuevo León
  - Instituto Nacional de Cancerologia, Distrito Federal
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, México
- Middlemore Clinical Trials, Auckland, New Zealand
- Peru (2):
  - Instituto Regional de Enfermedades Neoplásicas del Sur, Arequipa
  - Oncosalud Sac, Lima
- South Korea (6):
  - Pusan National University Hospital, Busan
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Yeouido St. Mary's Hospital, Seoul
- Thailand (4):
  - Chulalongkorn University Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai Uni Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen Uni, Khon Kaen
- Turkey (Türkiye) (4):
  - Ankara University Medical Faculty, Ankara
  - Medipol Mega Üniversite Hastanesi Göztepe, Istanbul
  - Anadolu Health Center, Kocaeli
  - Dokuz Eylul Universitesi Tip Fakultesi, Lzmir

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Budde LE, Zhang H, Kim WS, Maruyama D, Rego EM, Norasetthada L, Hong H, Ozcan M, Jeon YW, Leao Cordeiro de Farias D, Fogliatto LM, Pavlovsky A, Goto H, Olszewski AJ, Shah N, Hu B, Yin S, Wu H, To I, Ead WS, Ashby J, Janousek M, Pham S, Wang J, Kwan A, Batlevi CL, Wei MC, Westin J. Mosunetuzumab Plus Polatuzumab Vedotin in Transplant-Ineligible Refractory/Relapsed Large B-Cell Lymphoma: Primary Results of the Phase III SUNMO Trial. J Clin Oncol. 2025 Dec 20;43(36):3799-3811. doi: 10.1200/JCO-25-01957. Epub 2025 Oct 2. PMID 41037766